CLINICAL TRIAL: NCT00057525
Title: A Phase 1 Study of Safety and Immunogenicity of E. Coli-Derived Recombinant Protective Antigen (rPA), a New Anthrax Vaccine Administered by the Intramuscular (IM) Route in Healthy Adults
Brief Title: A New Anthrax Vaccine Administered by the Intramuscular (IM) Route in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DynPort Vaccine Company LLC, A GDIT Company (Industry)
Responsible Party: Chief Medical Officer, DynPort Vaccine Company, LLC
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: rPA-EC-02; Anthrax
Record Dates: First submitted 2003-04-03; First posted 2003-04-07 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Anthrax
Keywords: Anthrax
MeSH Terms: conditions — Anthrax | interventions — Charcoal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anthrax vaccine with or without PBS (Experimental): Administor 1 dose 5 μg rPA with PBS (5 Volunteers)
  Interventions: Biological: Anthrax
- Placebo (Placebo Comparator): Doses will range from 5 _g to 100 _g rPA, and at each dose-level, rPA will either be combinedwith phosphate-buffered saline (PBS) or adsorbed to Alhydrogel
  Interventions: Biological: Alhdryogel or PBS

INTERVENTIONS:
Biological: Anthrax — Doses will range from 5 _g to 100 _g rPA, and at each dose-level, rPA will either be combined with phosphate-buffered saline (PBS) or adsorbed to Alhydrogel
  Arms: Anthrax vaccine with or without PBS
Biological: Alhdryogel or PBS — Doses will range from 5 _g to 100 _g rPA, and at each dose-level, rPA will either be combined with phosphate-buffered saline (PBS) or adsorbed to Alhydrogel
  Arms: Placebo

SUMMARY:
This study will provide preliminary safety and comparative immunogenicity data for the E.coli derived rPA vaccine administered by intramuscular (IM) injection at Day 0 and Month 1.Doses will range from 5 μg to 100 μg rPA, and at each dose-level, rPA will either be combined with phosphate-buffered saline (PBS) or adsorbed to Alhydrogel.

DETAILED DESCRIPTION:
This is a safety study with an open-label part (2 groups), followed by a dose-ranging part evaluating safety and immunogenicity using a double-blind, sequential-group design with randomization and placebo-control within each of the 6 groups. Volunteers in each dose group will receive two IM injections at Day 0 and Month 1

ELIGIBILITY:
Volunteers are eligible for this study if they meet all the following criteria:

* Citizens of the U.S.
* Age 18 to 40 years.
* For women, a negative serum pregnancy test will be required at study entry and within 24 hours prior to each vaccination, as well as verbal assurance that adequate birth control measures are applied prior to initial vaccination and for 3 months after the last vaccination.
* Good health as determined by medical history, physical examination, and clinical judgment.
* Normal Baseline Clinical Laboratory Values at screening including:

  * Complete Blood Count (CBC) including:
  * White Blood Cell Count: 3.8 -10.8
  * Red Blood Cell Count (Mill/MCL)
  * Male: 4.20 - 5.80
  * Female: 3.80 - 5.10
  * Hemoglobin (G/DL)
  * Male: 13.2 - 17.1
  * Female: 11.7 - 15.5
  * Hematocrit (%)
  * Male: 38.5- 50.0
  * Female: 35.0 - 45.0
  * Platelet Count: 140 - 440 (THOUS/MCL)
  * Differential
  * Urine dipstick for protein and blood: negative or trace. If either is ≥ 1+, obtain complete urinalysis (UA). If microscopic UA confirms evidence of hematuria or proteinuria ≥ 1+, the volunteer is ineligible.
  * Negative serology for HIV infection (ELISA test).
  * CPK within normal limits
  * Hepatic Function Tests including AST, ALT, ALK PHOS.
  * Total bilirubin, BUN, serum creatinine, serum electrolytes
* Availability for at least 13 months of follow-up from the time of the screening visit.
* Successful completion of the Test of Understanding defined as 90% correct with three opportunities to take test. Errors will be reviewed with volunteer after each test.
* Commitment for trial participation and signature of the approved consent form.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2003-04; Primary Completion 2004-04 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merlin L Robb, MD, Principal Investigator — Walter Reed Army Institute of Research / Henry M. Jackson Foundation Vaccine Clinical Research Center, 1600 East Gude Dr., Rockville, MD 20850
Locations (1):
- Walter Reed Army Institute of Research / Henry M. Jackson Foundation Vaccine Clinical Research Center, 1600 East Gude Dr, Rockville, Maryland, United States

REFERENCES:
- [Derived] Brown BK, Cox J, Gillis A, VanCott TC, Marovich M, Milazzo M, Antonille TS, Wieczorek L, McKee KT Jr, Metcalfe K, Mallory RM, Birx D, Polonis VR, Robb ML. Phase I study of safety and immunogenicity of an Escherichia coli-derived recombinant protective antigen (rPA) vaccine to prevent anthrax in adults. PLoS One. 2010 Nov 5;5(11):e13849. doi: 10.1371/journal.pone.0013849. PMID 21079762